CLINICAL TRIAL: NCT00399620
Title: Chromogranin-A-Derived Peptides in the Gingival Crevicular Fluid and the Saliva of Diabetic Patients With or Without Periodontitis
Brief Title: Chromogranin-A-Derived Peptides and Periodontitis in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3739
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Periodontitis and Diabetitis
Keywords: Periodontitis; Diabetes; Gingival crevicular fluid; GCF; Saliva; Chromogranin; Electrophorèse; Western Blot; RT-HPLC
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Gingival crevicular fluid samples (this procedure is added to the subject usual medical follow-up).

SUMMARY:
Periodontitis is a chronic disease of the supporting tissue of the teeth, characterized by bleeding and inflamed gingival, resorption of alveolar bone. This disease has a significant impact of the quality of life as the teeth become progressively mobile and may fall out spontaneously if no treatment is provided. Periodontal disease has been cited as the sixth complication of diabetes mellitus.Chromogranins / secretogranins are a family of proteins present in nervous endocrine and immune cells, released with catecholamines during stress situations. Chromogranin A (CGA) is the major member of this family.The aim of this study is to determine the level of CGA and its derived peptides in the gingival crevicular fluid (GCF) of health or diabetic patients with and without periodontitis.Then, we want to determine the antimicrobial activity of these peptides.

ELIGIBILITY:
Inclusion criteria:

* Patients from 20 to 80 years old
* A minimum of 10 teeth
* Healthy volunteers or diabetic patients with or without periodontitis

Exclusion criteria:

* a course of antibiotics
* a fungicidal therapy
* a corticotherapy
* a hormone therapy
* a pregnancy
* persons under guardianship

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2008-03

CONTACTS AND LOCATIONS:
Overall Officials: Martine Soell, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Département de Parodontologie - Hôpital Civil, Strasbourg, France